CLINICAL TRIAL: NCT06646055
Title: A Phase Ib/II Clinical Study of AK112 and Cadonilimab Combined With Chemotherapy as First-line Treatment for Metastatic Pancreatic Cancer
Brief Title: AK112 and Cadonilimab Combined With Chemotherapy for 1L Treatment of Metastatic Pancreatic Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AK112-210
Record Dates: First submitted 2024-10-16; First posted 2024-10-17 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Metastatic Pancreatic Ductal Adenocarcinoma
MeSH Terms: interventions — 130-nm albumin-bound paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Cadonilimab(q4w) + AK112 + nab-paclitaxel + gemcitabine(phase Ib) (Experimental): Cadonilimab will be administered at a selected dose every 4 weeks (q4w). AK112 will be administed at a fixed dose every 2 weeks (q2w). Nab-paclitaxel and gemcitabine will be administed at 125mg/m2 d1, d8, d15 q4w, and 1000mg/m2 d1, d8, d15 q4w, intravenously respectively.
  Interventions: Drug: AK112, Cadonilimab, nab-paclitaxel, gemcitabine
- Cadonilimab(q2w) + AK112 + nab-paclitaxel + gemcitabine(phase Ib) (Experimental): Cadonilimab will be administered at a selected dose every 2 weeks (q2w). AK112 will be administed at a fixed dose every 2 weeks (q2w). Nab-paclitaxel and gemcitabine will be administed at 125mg/m2 d1, d8, d15 q4w, and 1000mg/m2 d1, d8, d15 q4w, intravenously respectively.
  Interventions: Drug: AK112, Cadonilimab, nab-paclitaxel, gemcitabine
- Cadonilimab + AK112 + nab-paclitaxel + gemcitabine(phase II) (Experimental): Cadonilimab will be administered at a selected dose and frequency from phase Ib. AK112 will be administered at a fixed dose every 2 weeks (q2w). Nab-paclitaxel and gemcitabine will be administed at 125mg/m2 d1, d8, d15 q4w, and 1000mg/m2 d1, d8, d15 q4w, intravenously respectively.
  Interventions: Drug: AK112, Cadonilimab, nab-paclitaxel, gemcitabine
- AK112 + nab-paclitaxel + gemcitabine(phase II) (Experimental): AK112 will be administered at a fixed dose every 2 weeks (q2w). Nab-paclitaxel and gemcitabine will be administed at 125mg/m2 d1, d8, d15 q4w, and 1000mg/m2 d1, d8, d15 q4w, intravenously respectively.
  Interventions: Drug: AK112, nab-paclitaxel, gemcitabine
- nab-paclitaxel + gemcitabine(phase II) (Active Comparator): Nab-paclitaxel and gemcitabine will be administed at 125mg/m2 d1, d8, d15 q4w, and 1000mg/m2 d1, d8, d15 q4w, intravenously respectively.
  Interventions: Drug: nab-paclitaxel, gemcitabine

INTERVENTIONS:
Drug: AK112, Cadonilimab, nab-paclitaxel, gemcitabine — IV infusion, specified dose on specified days.
  Arms: Cadonilimab(q4w) + AK112 + nab-paclitaxel + gemcitabine(phase Ib)
Drug: AK112, Cadonilimab, nab-paclitaxel, gemcitabine — IV infusion, specified dose on specified days.
  Arms: Cadonilimab(q2w) + AK112 + nab-paclitaxel + gemcitabine(phase Ib)
Drug: AK112, Cadonilimab, nab-paclitaxel, gemcitabine — IV infusion, specified dose on specified days.
  Arms: Cadonilimab + AK112 + nab-paclitaxel + gemcitabine(phase II)
Drug: AK112, nab-paclitaxel, gemcitabine — IV infusion, specified dose on specified days.
  Arms: AK112 + nab-paclitaxel + gemcitabine(phase II)
Drug: nab-paclitaxel, gemcitabine — IV infusion, specified dose on specified days.
  Arms: nab-paclitaxel + gemcitabine(phase II)

SUMMARY:
This trial is a Phase Ib/II study. All patients are stage IV pancreatic cancer (PDAC) patients with Eastern Cooperative Oncology Group (ECOG) performance status of 0-1. The purpose of this study is to evaluate the safety and efficacy of AK112 and Cadonilimab combined with chemotherapy as first-line treatment for patients with metastatic pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Be able and willing to provide written informed consent and to comply with all requirements of study participation (including all study procedures).
2. ≥18 years old and ≤ 75 years (regardless of sex).
3. ECOG performance status 0-1
4. Life expectancy longer than 3 months.
5. Histologically or cytologically confirmed diagnosis of metastatic pancreatic ductal carcinoma (PDAC).
6. No prior systemic anti-tumor therapy for metastatic PDAC.
7. Adequate organ function.
8. Measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.

Exclusion Criteria:

1. Histological or cytological diagnosis of other pathological types.
2. BRCA1/2 or PALB2 mutations.
3. Participating in another clinical research.
4. Active central nervous system (CNS) metastases.
5. Undergoing systemic antiangiogenic therapy.
6. Acute or subacute pancreatitis.
7. Other known malignancies within five years.
8. Active infection requiring systemic therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-01-21 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Frequency of adverse events (AEs) and serious adverse events (SAEs) | 28days+28days
  Frequency of AEs and SAEs for all Arms in phase Ib.
Overall Response Rate (ORR) | Up to approximately 2 years
  ORR is the proportion of subjects with complete response(CR) or partial response(PR) , based on RECIST v1.1.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) | Up to Cycle 12
  PK parameters: serum concentrations of AK112 and Cadonilimab at different point of time
Anti-Drug Antibodies(ADAs) | Up to approximately 2 years
  Number and percentage of patients with detectable anti-drug antibodies
Progression-Free Survival (PFS) | Up to approximately 2 years
  Evaluation of PFS based on RECIST v1.1.
Overall survival (OS) | Up to approximately 2 years
  Evaluation of OS based on RECIST v1.1.
Disease control rate (DCR) | Up to approximately 2 years
  Evaluation of DCR based on RECIST v1.1.
Duration of Response (DoR) | Up to approximately 2 years
  Evaluation of DoR based on RECIST v1.1.
Time to Response (TTR) | Up to approximately 2 years
  Evaluation of TTR based on RECIST v1.1.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science & Technology., Wuhan, Hubei, China